CLINICAL TRIAL: NCT02378831
Title: Testing for Sleep Apnea in Adolescence Subjects With the WP200/WP200U Compared to an In-lab Overnight PSG Testing
Brief Title: Comparison of In-lab PSG to WP200 for Assessing Sleep Parameters
Status: Withdrawn | Type: Observational
Why Stopped: has not begun yet.
Sponsor: Itamar-Medical, Israel (Industry)
Responsible Party: Sponsor
Other Study IDs: WP200/U-adolescence- 001
Record Dates: First submitted 2015-02-17; First posted 2015-03-04 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-02

CONDITIONS: Sleep
Keywords: diagnosing sleep

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PSG and WatchPAT200 in subjects age12-17: Adolescents refered to a sleep lab for sleep lab for full night PSG

SUMMARY:
The WP200 and/or WP200U will be compared with a PSG system which is a digital physiological recorder system, cleared for use for clinical sleep studies. The manual scoring of the PSG data, performed by a trained and authorized scorer, according to the AASM (American Academy of Sleep Medicine) guidelines, serves as a "gold standard" for all determinations of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12-17
* Subjects with a legal guardian that is able to read understand and sign the informed consent form
* Willing to sleep with the WP200/WP200U and PSG simultaneously in the sleep lab

Exclusion Criteria:

* Permanent pacemaker: atrial pacing or VVI without sinus rhythm.
* Use of one of the following medications: alpha blockers, short acting nitrates (less than 3 hours before the study)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will include adolescence subjects, age 12-17, referred to the clinical sleep laboratory for an overnight sleep study
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
sensitivity, specificity, obtained by the WP200/WP200U device automatic-computerized analysis as compared to the manual scoring of the PSG that is considered the "gold standard" | 1 night
correlation obtained by the WP200/WP200U device automatic-computerized analysis as compared to the manual scoring of the PSG that is considered the "gold standard" | 1 night
Agreement obtained by the WP200/WP200U device automatic-computerized analysis as compared to the manual scoring of the PSG that is considered the "gold standard" | 1 night